CLINICAL TRIAL: NCT06468488
Title: Impact of Drainless Donor Abdominal Site in Deep Inferior Epigastric Perforator (DIEP) Flap on Complications and Duration of Hospital Stay.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Felix Debruyn, Medical doctor in plastic surgery, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S68700
Record Dates: First submitted 2024-05-26; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Breast Reconstruction
Keywords: Breast reconstruction; DIEP; Drainless
MeSH Terms: interventions — Drainage

STUDY DESIGN:
Intervention Model Description: Non blindend randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIEP flap surgery with drains (Active Comparator): Patients will undergo a breast reconstruction by a DIEP flap with drains.
  Interventions: Procedure: DIEP flap surgery with drains
- DIEP flap surgery without drains (Experimental): Patients will undergo a breast reconstruction by a DIEP flap without drains.
  Interventions: Procedure: DIEP flap surgery without drain

INTERVENTIONS:
Procedure: DIEP flap surgery without drain — Patients will undergo a breast reconstruction with a DIEP flap without the placement of drains.
  Arms: DIEP flap surgery without drains
Procedure: DIEP flap surgery with drains — Patients will undergo a breast reconstruction with a DIEP flap with the placement of drains.
  Arms: DIEP flap surgery with drains

SUMMARY:
Inserting surgical drains is an ancient approach used across different specialties because of its many advantages such as discharge of fluid accumulation, appraising and qualifying drain capacities, lowering infection percentages, and eliminating dead space.

Most commonly, abdominal closed-suction drains are used following autologous breast reconstruction with a DIEP flap to prevent donor site complications such as seroma, hematoma, and wound dehiscence. Although abdominal drains are effective in impeding accumulation, they are a potential portal for infection, Furthermore, they restrict patient mobility, are cumbersome, require time-consuming care upon discharge, potentially increase inpatient stay and ultimately resulting in impaired health-care costs. In the context of an Enhanced Rapid Protocol (ERP), not placing abdominal drains would be a step forward. This involves using "quilting sutures" to close the dead space after flap prelevation. Quilting sutures are placed between the subcutaneous tissues of the abdominal flap and the underlying fascia of the rectus abdominis muscle and aim to minimizes the shearing forces and collapse the death space without the use of drains. Progressive tension sutures were first described in 2000, in a retrospective paper on cosmetic abdominoplasty patients. Since then, their procedure has been analysed and adapted by many authors and applied in perforator-based abdominal flaps for breast reconstruction.

Despite the drainless approach is well known in the literature for cosmetic abdominoplasty procedures, prospective clinical investigations to encourage the drainless approach in DIEP flap reconstruction is lacking. Therefore we want to set up a prospective study to make a comparison between the outcomes succeeding donor site closure after DIEP flap harvesting with (AD) or without (W-AD) the use of abdominal drains and investigate whether there is a correlation between the use of drains and the length of hospital stay. Secondary outcomes involve the complication rate of seroma, hematoma, and dehiscence analysis of abdominal drain output and postoperative recovery, including pain and follow-up complications as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any screening procedures
2. Gender: female
3. Age >18 years old
4. Breast cancer for which mastectomy is planned (primary case) OR patient has already had mastectomy (secondary case)
5. Wish to have a DIEP flap procedure (uni-or bilateral) for breast reconstruction
6. Meets criteria for DIEP flap procedure (no previous open abdominal surgery)
7. Pre- and postoperative smoking cessation of 3 months

Exclusion Criteria:

1. Patient has history of open abdominal surgery wich compromises blood flow to DIEP flap
2. Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the CIP.
3. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method.
4. No informed consent
5. Age < 18 years old
6. Currently smoking or cessation <3 months preoperatively
7. The use of immunosuppressive drugs
8. Other ongoing therapies which might compromise normal postoperative course (e.g. chemotherapy, radiotherapy, …)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Length of stay (LOS) | During admission to the hospital
  Length of hospital stay (LOS) is the same or less in patients without abdominal drains versus patients with drains

SECONDARY OUTCOMES:
Complication rate | from enrollment until study completion, an average of 1 year
  Complications (hematoma, seroma, wound dehiscence, wound infection) are the same or less in patients without abdominal drains versus patients with drains
Pain (VAS) | from enrollment until study completion, an average of 1 year
  We will investigate if pain is the same or less in patiens without abdominal drains versus patients with drains. We will use the VAS (visual analogue scale)
Patient satisfaction (Breast Q) | from enrollment until study completion, an average of 1 year
  We will investigate if patient satisfaction is the same or less in patients without abdominal drains versus patients with drains. We will use the breast Q queestionnaire..

CONTACTS AND LOCATIONS:
Locations (1):
- Uz Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided